CLINICAL TRIAL: NCT02705794
Title: Clinical Trial of Comparative Evaluation of Modified Mallampati Score and Modified Mallampati Score Along With Thyromental Distance, Anatomical Abnormalities and Cervical Mobility in Predicting Difficult Airway
Brief Title: Comparison of Modified Mallampati Classification With M-TAC in Difficult Airway
Status: Completed | Type: Observational
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Bikramjit Das, Assistant Professor, Government Medical College, Haldwani
Other Study IDs: 124-IEC/01/13
Record Dates: First submitted 2016-02-11; First posted 2016-03-11 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Airway Management
Keywords: intubation, laryngoscopy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study title "Clinical trial of comparative evaluation of the Modified Mallampati Score and Modified Mallampati Score along with Thyromental distance, Anatomical abnormality, and Cervical mobility (M-TAC) in Predicting Difficult Airway " was undertaken to evaluate prediction of difficult airway by comparing preoperative airway evaluation tests.

Mallampati classification is the most used screening test for detection of difficult intubation it is a classification of oropharyngeal view. Other tests include sternomental distance, thyromental distance, Wilson risk sum score, upper lip bite test, protrusion of mandible, tooth morphology, head extension, mouth opening, body mass index, 3-3-2 rule and ultrasonography of neck soft tissue. We studied 200 adult ASA I & II patients of either sex, aged between 18-60 yrs undergoing elective surgery receiving general anesthesia.

Modified mallampati classification had four grades & each grade was given a score, similarly thyromental distance (TMD), anatomical abnormality (AA) & cervical mobility (CM) was classified into three grades & each grade was given a score. For M-TAC individual scores were added.

DETAILED DESCRIPTION:
The term 'airway' refers to the upper airway which may be defined as the extra-pulmonary air passage, consisting of the nasal and oral cavities, pharynx, larynx, trachea and large bronchi.

The most commonly applied methods of oxygenation is ventilation through a tracheal tube, a laryngeal mask, or a face mask. Problems with tracheal intubation remain the major cause of death and disability due to anaesthesia in analyses of records of the United Kingdom medical defence societies and in the American Society of Anaesthesiologists closed claims database.

'Difficult airway' is one in which there is a problem in establishing or maintaining gas exchange via a mask, an artificial airway or both. Prediction of difficult airway management remains a pivotal challenge for anaesthesiologists because accurate prediction gets altered the potentially dangerous unanticipated airway to an anticipated difficult airway with, predominantly, ample time for proper preparation. This is helpful in reducing potential complications by the allocation of experienced personnel and by using relevant equipment and well planned strategies .

However rare, in spite of this, occurrence of difficult airway management still occurs and it prompts to increase the risk of morbidity and mortality - especially when not anticipated. Unanticipated difficulty in intubation in patients for elective surgical procedures can occur in 1.5 to 13 percent cases with none of the above mentioned abnormalities resulting in both morbidity and mortality.

Several pre-operative risk factors for assessing airway difficulties have been identified, yet none have convincing diagnostic accuracy when using in isolation. Combining several risk factors increase the predictive value of the test and multivariable risk models have been developed.

As the anatomy of the head and neck region plays a leading role in deciding the fateful profile of the airway, especially associated with influential abnormality. So, simple bedside test, such as the modified Mallampati test, has been found to be of limited value and cannot be relied on for using in predicting difficult laryngoscopy. Exclusively when each individual was investigated in isolation using a single scoring test, as it has long been realized that difficult laryngoscopy is a multifactorial problem. Thus, effective prediction requires a combination of multiple tests to provide a high index of sensitivity and specificity for prediction of difficult airway. Thus, we ventured to combine Mallampati score with some other anatomical factors (thyromental distance, anatomical abnormality and cervical mobility) to develop a new and simpler clinical prediction model for a better predictive ability.

ELIGIBILITY:
Inclusion Criteria:

* -Adult patients aged 18-60 years.
* American Society of Anesthesiologists (ASA) I or II, scheduled for elective surgeries under general anaesthesia requiring endotracheal intubation

Exclusion Criteria:

* - Patient refusal
* ASA grade III and IV
* Cervical spine disorder
* Obstructive airway tumor
* Edentulous patients /Irregular dentition
* past history of difficult laryngoscopy and intubation.
* trauma to the airways or to the cranial, cervical, and facial regions
* history of previous surgery, burns to airways & adjacent structures
* Mouth opening<3 cm
* Age <18 years & > 60 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient admitted for various surgeries requiring general anesthesia with tracheal intubation in a tertiary care teaching institute
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Difficulty of intubation | 10 minutes
  Difficulty of intubation is assessed by modified Cormack and Lehane grading. Modified Cormack and Lehane and grading consists of 4 grades. Grade 3 and 4 is considered as difficulty intubation.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ambesh SP, Singh N, Rao PB, Gupta D, Singh PK, Singh U. A combination of the modified Mallampati score, thyromental distance, anatomical abnormality, and cervical mobility (M-TAC) predicts difficult laryngoscopy better than Mallampati classification. Acta Anaesthesiol Taiwan. 2013 Jun;51(2):58-62. doi: 10.1016/j.aat.2013.06.005. Epub 2013 Jul 21. PMID 23968655
- [Background] Khan ZH, Mohammadi M, Rasouli MR, Farrokhnia F, Khan RH. The diagnostic value of the upper lip bite test combined with sternomental distance, thyromental distance, and interincisor distance for prediction of easy laryngoscopy and intubation: a prospective study. Anesth Analg. 2009 Sep;109(3):822-4. doi: 10.1213/ane.0b013e3181af7f0d. PMID 19690252